Official title: Mindfulness-Based Intervention for Caregivers of Frail older adults: Towards a model of intergenerational caregiving for Chinese families

NCT number: to be assigned

Document date: April 22, 2021



## **Consent to Participate in Research**

## Family Psychoeducation Programme for Caregivers of Frail Older Adults

| | nsent to participate in the captioned research conducted by I<br>Department of Applied Social Sciences, The Hong Kor |
|---|---|
| Polytechnic University. | , Department of Applied Social Sciences, The Hong Kol |
| | ned from this research may be used in future research arrivacy will be retained, i.e. my personal details will not be |
| 1 | hed information sheet has been fully explained. I understandarticipation in the project is voluntary. |
| I acknowledge that I have the right t time without penalty of any kind. | o question any part of the procedure and can withdraw at an |
| Name of Participant | |
| Signature of Participant | |
| Name of Principal Investigator | Dr. Hay Ming LO |
| Signature of Principal Investigator | |
| Date | |